CLINICAL TRIAL: NCT04804800
Title: Virtual Reality Place in the Management of Body Dysmorphia Disorders in Anorexia Nervosa : Comparison of the Recommended Management and Virtual Reality Care Programs With or Without Multisensory Remedy
Brief Title: Virtual Reality Place in the Management of Body Dysmorphia Disorders in Anorexia Nervosa
Acronym: PROSANOR
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Lille Catholic University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: RC-P0089
Record Dates: First submitted 2021-03-16; First posted 2021-03-18 (Actual); Last update posted 2022-01-06 (Actual); Status verified 2022-01

CONDITIONS: Anorexia Nervosa; Dysmorphophobia
Keywords: Anorexia Nervosa; Dysmorphophobia; Body distortions; Multisensory remediation; Virtual Reality
MeSH Terms: conditions — Anorexia Nervosa; Body Dysmorphic Disorders

STUDY DESIGN:
Intervention Model Description: This study presents three groups of patients :
  * The control group : The patients benefit from the care recommended by the HAS, relaxation times and body scan.
  * The experimental group 1 : The patients benefit from the care recommended by the HAS, the virtual reality program and relaxation times and body scan.
  * The experimental group 2 : The patients benefit from the care recommended by the HAS, the virtual reality program, the multi-sensory remediation and relaxation times and body scan.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control group (No Intervention): The patients benefit from the care recommended by the HAS. They benefit from psychological interviews, psychiatric follow-up, dietetic follow-up, family interviews and therapy. Body therapies (physiotherapy, massage, fascia therapy, psychomotor skills, dance therapy, etc.) may also take place. Patients will also benefit from relaxation and body scan.
- Experimental group 1 : Virtual Reality (Experimental): The patients benefit from the care recommended by the HAS, the virtual reality program and time for relaxation and body scan (1 hour).
  Interventions: Other: Experimental group 1 : Virtual Reality
- Experimental group 2 : Virtual Reality + Multi Sensorial Remediation (Experimental): The patients benefit from the care recommended by the HAS, the virtual reality and the multisensory remediation programs, and also the body scan.
  Interventions: Other: Experimental group 2 : Virtual Reality + Multi Sensorial Remediation

INTERVENTIONS:
Other: Experimental group 1 : Virtual Reality — Patients benefit from the care recommended by the HAS, the virtual reality program and time for relaxation and body scan.
  Arms: Experimental group 1 : Virtual Reality
Other: Experimental group 2 : Virtual Reality + Multi Sensorial Remediation — Patients benefit from the care recommended by the HAS, the virtual reality program, the multisensory remediation, and also the body scan.
  Arms: Experimental group 2 : Virtual Reality + Multi Sensorial Remediation

SUMMARY:
Body distortions are responsible for anorexic behavior reinforcing loops. It is necessary to target this behavior and develop appropriate therapies taking into account the perceptual (implicit) and conceptual (explicit) phenomenon of body representations.

The main originality of the proposed program consists on combining virtual visual impulses and multisensory recalibration (touch, proprioception, vestibular sensations) in order to compare the body distortions evolution in anorexic patients with or without a multimodal care program including Virtual Reality from its own body scan, coupled or not to a multisensory remediation.

DETAILED DESCRIPTION:
Rapid weight loss associated with mental anorexia leads to dysmorphophobia and body distortions. Patients perceive themselves to be bigger than they really are. Body distortions are responsible for anorexic behavior reinforcing loops. It is then necessary to target this behavior and develop appropriate therapies taking into account the perceptual (implicit) and conceptual (explicit) phenomenon of body representations.

The current treatment programs which are recommended by the Haute Autorité de Santé (HAS) in France focus on the somatic, nutritional, individual and family psychological aspects. These recommendations hardly mention the bodily distortion phenomenon which frequently leads patients to relapse into the disease.

The 3D body scanner enables to get awareness of the body through visual feedback allowing the patient to get a reassuring overview of her weight development.

This projects aims to combine virtual visual impulses and multisensory recalibration (touch, proprioception, vestibular sensations) in order to compare the body distortions evolution in anorexic patients with or without a multimodal care program including Virtual Reality from its own body scan coupled or not to a multisensory remediation.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Age ≥ 15 to ≤ 26 years old
* Anorexic nervosa eating disorder according to the criteria of Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM 5). As patients are hospitalized for anorexic nervosa, the medical diagnosis of each care center participating in the inclusions will be trusted
* Patient hospitalized (full hospitalization or day hospital) in one of the investigative centers for a minimum period of 6 weeks
* 14 ≤ BMI ≤ 18.5 for adult patients. For minors, Cole's curves will be used. The Body mass index (BM)I should be between the 1st percentile and the 10th percentile (if the weight curve shows a clear break indicating abnormal weight loss). For example, for a 15-year-old girl, the BMI should be between 14.5 and 16.8.
* Presence of body distortion (BSC ≥ 20%)
* French language mastery
* Affiliation to a social security system
* Signature of informed consent to participate in this study by the patient and by her parents in the case of underage patients

Exclusion Criteria:

* Associated major mental disorders (psychotic disorders, bipolar disorders, major depression)
* Neurological disorders (pyramidal or extrapyramidal syndromes)
* Substance addiction (drugs, alcohol)
* Any disorder likely to impair the reasoning, discernment or judgment abilities
* Psychological incapacity to answer the questionnaires
* Medical contraindication to the practice of physical activity (identical contraindication to people without anorexia. In fact, appropriate physical activity is prescribed in anorexic patients in order to reduce the cardiovascular risks, osteopenia or anxiety and allow them to become aware of an adapted physical practice (reduction of anarchic physical hyperactivity)
* Participation in other research programs or psychomotor treatments in parallel
* Pregnant or breastfeeding woman
* Persons under guardianship, curatorship or legal protection
* Blindness, eye infections, mask wounds, poorly balanced epilepsy, psychiatric disorders incompatible with virtual reality

Ages: 15 Years to 26 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 150 (Estimated)
Dates: Start 2022-09 (Estimated); Primary Completion 2025-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Change in Body Dimensions Estimation task | 6 weeks
  Body overestimation bias will be assessed by the Body Dimensions Estimation task.

SECONDARY OUTCOMES:
Change in Body Shape Questionnaire | 6 weeks
  The womens body image concerns will be evaluated by the Body Shape Questionnaire. This 34-items questionnaire is scored from 1 (= never) to 6 (= always) to obtain a global score.
Change in Physical self description questionnaire | 6 weeks
  The Physical self description will be measured by the Physical Self Description Questionnaire (PSQD). This questionnaire estimates 11 sub-dimensions of the physical self from 70 items on a continuum ranging from 1 (very negative perception) to 6 (very positive perception).
Change in Body Image Questionnaire | 6 weeks
  Patients bodily satisfaction will be assessed by the Body Image Questionnaire. This questionnaire consists of 19 items scored on 5 points. It gives a total body satisfaction score between 19 and 95 and 4 scores relative to 4 different factors (accessibility/closure, satisfaction/dissatisfaction, active/passive, serenity/tension).
Change in Weight gain | 6 weeks
  Weight gain will be measured by weighting.
Change in Eating Disorder Examination Questionnaire | 6 weeks
  Eating disorders will be assessed by the Eating Disorder Examination Questionnaire (EDE-Q). This questionnaire is divided into several sub-scores: restriction, dietary concerns, body shape concerns and weight concerns. It has 30 items scored from 0 (= no day) to 6 (= every day). A score for each subscale and an overall score can be obtained.
Anxiety measured by the State-Trait Anxiety Inventory (STAI-Etat-Trait) | 6 weeks
  Anxiety will be measured by the STAI-Etat-Trait . Each of the dimensions (STAI-state and Stai-trait) are measured by 20 items scored from 1 (= no or never) to 4 (= yes or almost always) which is summarized by a score.

CONTACTS AND LOCATIONS:
Overall Officials: Vincent Dodin, PhD, Principal Investigator — Hôpital Saint-Vincent de Paul

IPD SHARING:
Plan to Share IPD: No